CLINICAL TRIAL: NCT05142189
Title: LuCa-MERIT-1: First-in-human, Open Label, Phase I Dose Confirmation Trial Evaluating the Safety, Tolerability and Preliminary Efficacy of BNT116 Alone and in Combinations in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Clinical Trial Evaluating the Safety, Tolerability and Preliminary Efficacy of BNT116 Alone and in Combinations in Patients With Advanced Non-small Cell Lung Cancer
Acronym: LuCa-MERIT-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BNT116-01; 2021-004739-94 (EudraCT Number); 2023-509283-14-00 (EU CTIS Number)
Record Dates: First submitted 2021-11-24; First posted 2021-12-02 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Cancer Vaccine; Non-Small Cell Lung Cancer; Combination with chemotherapy; Combination with other investigational agents; anti-cytotoxic T-lymphocyte-associated protein 4 [CTLA-4] antibody; anti-B7-H3 antibody conjugated to topoisomerase I inhibitor; anti-HER3 antibody conjugated to topoisomerase I inhibitor; Immunotherapy; Antibody-drug conjugate (ADC); Combination with a PD-1 inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cemiplimab; Docetaxel; Carboplatin; Paclitaxel; Antibodies, Bispecific; Vascular Endothelial Growth Factor A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Cohort 1A - BNT116 Monotherapy (Experimental)
  Interventions: Biological: BNT116
- Cohort 1B - BNT116 Monotherapy (Experimental)
  Interventions: Biological: BNT116
- Cohort 2 - BNT116 + Cemiplimab (PD-1/PD-L1 Inhibitor Refractory/Relapsed Participants) (Experimental)
  Interventions: Biological: BNT116; Biological: Cemiplimab
- Cohort 3 - BNT116 + Docetaxel (Experimental)
  Interventions: Biological: BNT116; Drug: Docetaxel
- Cohort 4 - BNT116 + Cemiplimab (Frail Participants) (Experimental)
  Interventions: Biological: BNT116; Biological: Cemiplimab
- Cohort 5 - BNT116 + Cemiplimab (After Concurrent Chemoradiotherapy [CRT]) (Experimental)
  Interventions: Biological: BNT116; Biological: Cemiplimab
- Cohort 6 - BNT116 + Cemiplimab + Carboplatin + Paclitaxel (Experimental): BNT116 + cemiplimab + carboplatin + paclitaxel as neo-adjuvant treatment followed by surgery, thereafter adjuvant treatment with BNT116 + cemiplimab
  Interventions: Biological: BNT116; Biological: Cemiplimab; Drug: Carboplatin; Drug: Paclitaxel
- Cohort 7 - BNT116 + BNT316 (Experimental): Dose finding for the combination of BNT116 with BNT316 (CTLA4 antibody) with dose escalation of BNT316
  Interventions: Biological: BNT116; Biological: BNT316
- Cohort 8: BNT116 + Anti-B7-H3 Antibody Conjugated to Topoisomerase I Inhibitor (Experimental): Dose finding for the combination of BNT116 with an anti-B7-H3 antibody conjugated to a topoisomerase I inhibitor with dose escalation of the anti-B7-H3 antibody conjugated to a topoisomerase I inhibitor
  Interventions: Biological: BNT116; Biological: anti-B7-H3 antibody conjugated to topoisomerase I inhibitor
- Cohort 9: BNT116 + Anti-HER3 Antibody Conjugated to Topoisomerase I Inhibitor (Experimental): Dose confirmation for the combination of BNT116 with an anti-HER3 antibody conjugated to a topoisomerase I inhibitor with dose escalation of the anti-HER3 antibody conjugated to a topoisomerase I inhibitor
  Interventions: Biological: BNT116; Biological: anti-HER3 antibody conjugated to topoisomerase I inhibitor
- Cohort 10: BNT116 + Bispecific Antibody for PD-L1 and VEGF-A (Frail Participants) (Experimental): Dose confirmation for BNT116 in combination with a bispecific antibody for programmed death ligand 1 (PD-L1) and vascular endothelial growth factor A (VEGF-A) will be established.
  Interventions: Biological: BNT116; Biological: Bispecific antibody for PD-L1 and VEGF-A
- Cohort 11: BNT116 + Bispecific Antibody for PD-L1 and VEGF-A (After Concurrent CRT) (Experimental): Dose confirmation for BNT116 in combination with a bispecific antibody for PD-L1 and VEGF-A will be established in participants after concurrent CRT.
  Interventions: Biological: BNT116; Biological: Bispecific antibody for PD-L1 and VEGF-A

INTERVENTIONS:
Biological: BNT116 — Intravenous injection
Biological: Cemiplimab — Intravenous infusion
  Arms: Cohort 2 - BNT116 + Cemiplimab (PD-1/PD-L1 Inhibitor Refractory/Relapsed Participants); Cohort 4 - BNT116 + Cemiplimab (Frail Participants); Cohort 5 - BNT116 + Cemiplimab (After Concurrent Chemoradiotherapy [CRT]); Cohort 6 - BNT116 + Cemiplimab + Carboplatin + Paclitaxel
Drug: Docetaxel — Intravenous infusion
  Arms: Cohort 3 - BNT116 + Docetaxel
Drug: Carboplatin — Intravenous infusion
  Arms: Cohort 6 - BNT116 + Cemiplimab + Carboplatin + Paclitaxel
Drug: Paclitaxel — Intravenous infusion
  Arms: Cohort 6 - BNT116 + Cemiplimab + Carboplatin + Paclitaxel
Biological: BNT316 — Intravenous infusion
  Arms: Cohort 7 - BNT116 + BNT316
Biological: anti-B7-H3 antibody conjugated to topoisomerase I inhibitor — Intravenous infusion
  Arms: Cohort 8: BNT116 + Anti-B7-H3 Antibody Conjugated to Topoisomerase I Inhibitor
Biological: anti-HER3 antibody conjugated to topoisomerase I inhibitor — Intravenous infusion
  Arms: Cohort 9: BNT116 + Anti-HER3 Antibody Conjugated to Topoisomerase I Inhibitor
Biological: Bispecific antibody for PD-L1 and VEGF-A — Intravenous infusion
  Arms: Cohort 10: BNT116 + Bispecific Antibody for PD-L1 and VEGF-A (Frail Participants); Cohort 11: BNT116 + Bispecific Antibody for PD-L1 and VEGF-A (After Concurrent CRT)

SUMMARY:
This first-in-human (FIH) trial for BNT116 aims to establish the safety profile and a safe dose for BNT116 monotherapy as well as for BNT116 in combination with approved medicinal products and/or in combination with investigational medicinal products (IMPs) including, but not limited to, cemiplimab, docetaxel, carboplatin, paclitaxel, BNT316 (an anti-cytotoxic T-lymphocyte-associated protein 4 [CTLA-4] antibody), an anti-B7-H3 antibody conjugated to a topoisomerase I inhibitor, an anti-human epidermal growth factor receptor 3 (HER3) antibody conjugated to a topoisomerase I inhibitor or a bispecific antibody for programmed death ligand 1 (PD-L1) and vascular endothelial growth factor A (VEGF-A) in participants with non-small cell lung cancer (NSCLC).

The trial will comprise of several cohorts for dose confirmation in monotherapy as well as in combinations of BNT116 as mentioned above.

The trial will enroll participants with NSCLC in advanced or metastatic stage in Cohorts 1 to 4 and Cohorts 7 to 10, unresectable NSCLC Stage III in Cohorts 5 and 11, and resectable NSCLC of Stage II and III in Cohort 6.

DETAILED DESCRIPTION:
The maximum duration of treatment for each individual participant in this trial is:

* Cohorts 1 to 4, and Cohorts 7 to 10: 24 months
* Cohorts 5 and 11: 18 cycles, i.e., 12 months
* Cohort 6: 4 cycles of neo-adjuvant treatment and 18 cycles of adjuvant treatment, i.e., 12 months of adjuvant treatment

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must have histologically confirmed NSCLC and measurable disease by RECIST v1.1. Note: Participants in Cohorts 1, 5 and 11 do not have to present with measurable disease.

  1. Participants must present with unresectable Stage III or metastatic Stage IV NSCLC by American Joint Commission on Cancer (AJCC) Cancer Staging Manual, Eighth Edition.

     EXCEPT
  2. Participants in Cohorts 5 and 11 must present with unresectable Stage III NSCLC by AJCC Cancer Staging Manual, Eighth Edition before receiving pre-trial chemoradiotherapy.
  3. Participants in Cohort 6 with the initial diagnosis of resectable Stage II and Stage III NSCLC by AJCC Cancer Staging Manual, Eighth Edition.
* Participants in Cohorts 2, 4, 5, 6, 10 and 11 must be able to tolerate (additional) anti-PD-1 therapy (i.e., did not permanently discontinue anti-programmed death protein 1 [PD-1] / programmed death ligand 1 [PD-L1] therapy due to toxicity).
* Participants must have an Eastern Cooperative Oncology Group performance status (ECOG-PS) less than or equal to (<=) 1, except for participants in Cohorts 1, 4, 5, 10 and 11 who are eligible with an ECOG-PS of 0-2.

Cohort-specific inclusion criteria:

Cohort 1:

* Participants prior therapy must have included at least a PD-1/PD-L1 inhibitor and a platinum-based chemotherapy regimen as well as one other line of systemic therapy (except if a participant is not candidate for a platinum-based chemotherapy and/or PD-1/PD-L1 inhibitor and/or another line of systemic therapy). Note: Participants newly enrolled in Cohort 1B under protocol v 5.0 and subsequent versions of the protocol must consent to mandatory blood sampling for peripheral blood mononuclear cells (PBMCs).
* Participants who are to start cemiplimab at Cycle 3 must present with PD-L1 expression of tumor proportion score (TPS) greater than or equal to (>=) 1% in tumor cells (as determined locally).

Cohort 2:

* Participants must present with PD-L1 expression of tumor proportion score (TPS) >= 50% in tumor cells (as determined locally prior to inclusion in this trial).
* Participants must present with progressive disease either

  1. in the advanced or metastasized stage of NSCLC: while on a PD-1/PD-L1 inhibitor therapy or within 6 months of termination of this treatment as first-line treatment. Or
  2. be refractory to ongoing adjuvant therapy/maintenance treatment after CRT with a PD-1/PD-L1 inhibitor that has been given for at least 3 months in monotherapy (i.e., after an initial combination therapy) before being enrolled into this trial.

Cohort 3:

* Participants prior therapy must have included at least a PD-1/PD-L1 inhibitor and a platinum-based chemotherapy regimen (except if a participant is not candidate for a platinum-based chemotherapy and/or PD-1/PD-L1 inhibitor).
* Participants must present with progressive disease.

Cohort 4:

* Participants who are not candidates for chemotherapy as first-line treatment for the advanced or metastasized stage of NSCLC may be enrolled if presenting with PD-L1 expression: TPS >= 1% in tumor cells (as determined locally).

Cohort 5:

* Participants NSCLC must have been considered unresectable due to participant's condition and/or tumor-related factors and the participants must have undergone chemoradiotherapy before entering the trial.

Cohort 6:

* Participants NSCLC must be considered technically and medically resectable.
* Participants must be considered eligible for neo-adjuvant treatment.

Cohort 7:

* Participants prior therapy must have included at least a PD-1/PD-L1 inhibitor and a platinum-based chemotherapy regimen (except if a participant is not a candidate for a platinum-based chemotherapy and/or PD-1/PD-L1 inhibitor). Note 1: Participants may have received prior therapy targeting CTLA-4, lymphocyte-activation gene 3 (LAG-3), T cell immunoglobulin and immunoreceptor tyrosine-based inhibitory motif [ITIM] domain (TIGIT), VEGF or VEGF receptor (VEGFR) inhibitor as monotherapy or part of a combination therapy. Note 2: If the participants' prior therapies included a CTLA-4 inhibitor, the participant must be able to tolerate (additional) treatment with the CTLA-4 inhibitor.
* Participants must present with progressive disease at trial enrollment.
* Participants must consent to mandatory blood sampling for PBMCs.

Cohorts 8 & 9:

* Participants prior therapy must have included at least a PD-1/PD-L1 inhibitor and a platinum-based chemotherapy regimen (except if a participant is not a candidate for a platinum-based chemotherapy and/or PD-1/PD-L1 inhibitor).
* Participants must present with progressive disease at trial enrollment.

Cohort 10:

* Participants who are not candidates for chemotherapy as first-line treatment for the advanced or metastasized stage of NSCLC may be enrolled.

Cohort 11:

* Participant's NSCLC must have been considered unresectable due to participants condition and/or tumor related factors and the participants must have undergone chemoradiotherapy before entering the trial.

Key Exclusion Criteria:

* Ongoing active systemic treatment against NSCLC.
* Presence of a driver mutation for which approved target therapies are available except if the participant is not a candidate for the respective targeted therapy.
* Ongoing or recent evidence (within the last 5 years) of significant autoimmune disease that required treatment with systemic immunosuppressive treatments which may suggest risk for immune-related adverse events. Note: Participants with autoimmune-related hyperthyroidism, autoimmune-related hypothyroidism who are in remission, or on a stable dose of thyroid-replacement hormone, vitiligo, or psoriasis may be included.
* Current evidence of new or growing brain or spinal metastases during screening. Participants with leptomeningeal disease are excluded. Participants with known brain or spinal metastases may be eligible for all Cohorts, except for Cohorts 5, 6 and 11, if they:
* had radiotherapy or another appropriate therapy for the brain or spinal metastases, AND
* have no neurological symptoms that can be attributed to the current brain lesions, AND
* have stable brain or spinal disease on the computed tomography (CT) or magnetic resonance imaging (MRI) scan within 4 weeks before signing the informed consent (confirmed by stable lesions on two scans at least 4 weeks apart), AND
* do not require steroid therapy for the treatment of brain or spinal metastases within 14 d before the first dose of trial treatment. Note: Spinal bone metastases (that is, of the vertebrae) are allowed, unless imminent fracture or cord compression is anticipated.
* Systemic immune suppression:
* Current use of chronic systemic steroid medication (<= 5 mg/day prednisolone equivalent is allowed); participants using physiological replacement doses of prednisone for adrenal or pituitary insufficiency are eligible. Note: Steroid medication given for supportive or prophylactic reasons during CRT for participants in Cohorts 5 and 11 needs to be tapered to <= 5 mg/day prednisolone equivalent at latest on the day before the trial treatment starts.
* Other clinically relevant systemic immune suppression within the last 3 months before trial enrollment.
* Known history of seropositivity for human immunodeficiency virus (HIV) with CD4+ T-cell (CD4+) counts less than (<) 350 cells/microlitre (mcL) and with a history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections.
* Prior splenectomy.
* History/risk of interstitial lung disease or low baseline lung function (baseline pulse oximetry of less than 92% oxygen saturation [SpO2] without additional oxygen).

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply to all or some participants depending on the cohort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Cohorts 1, 2, 3, 4, 6, 7, 8, 9, 10 and 11: Occurrence of Dose-Limiting Toxicities (DLTs) During the DLT Observation Period | From first dose of IMP up to 21 days
Cohorts 1 to 11: Occurrence of Treatment-Emergent Adverse Events (TEAEs) Reported by Relationship, Seriousness, and Grade | up to 27 months
  According to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0
Cohort 6 only: Occurrence of Post-Surgical Adverse Events (AEs) Related to BNT116 and Cemiplimab | up to 27 months
Cohort 6 only: Occurrence of Treatment-Related Delays to Surgery More Than 9 weeks Post the Last Dose of Neo-Adjuvant Treatment | up to 6 months

SECONDARY OUTCOMES:
Cohorts 1, 2, 3, 4, 7, 8, 9, and 10: Overall Response Rate (ORR) | up to 27 months
  ORR defined as the number of participants with complete response (CR) or partial response (PR) as best overall response (BOR) according to response evaluation criteria in solid tumors (RECIST) v1.1 divided by the number of patients in the efficacy analysis set.
Cohorts 1, 2, 3, 4, 7, 8, 9, and 10: Duration of Response (DoR) | up to 27 months
  DoR defined as the time from initial response until first objective tumor progression according to RECIST v1.1.
Cohorts 1, 2, 3, 4, 7, 8, 9, and 10: Disease Control Rate (DCR) | up to 27 months
  DCR defined as the number of participants with CR or PR or stable disease (SD) as BOR according to RECIST v1.1 divided by the number of patients in the efficacy analysis set.
Cohorts 1, 2, 3, 4, 7, 8, 9, and 10: Duration of Disease Control | up to 27 months
  Duration of disease control defined as the time from initial detection of stable disease or response until first objective tumor progression according to RECIST v1.1.
Cohorts 1, 2, 3, 4, 7, 8, 9, and 10: Progression-Free Survival (PFS) | up to 48 months
  PFS defined as the time of first trial treatment until the first objective tumor progression according to RECIST v1.1 or death from any cause, whichever occurs first.
All cohorts: Overall Survival (OS) | up to 48 months
  OS defined as the time of first trial treatment until death from any cause.
Cohort 5, 6 and 11: Event Free Survival (EFS) | up to 48 months
  EFS defined as the length of time from first trial treatment to any of the following events: progression of disease, recurrence of disease or death from any cause, whichever occurs first.
Cohort 5, 6 and 11: EFS Rate at 12 and 24 months | up to 24 months
  EFS rate defined as the number of participants without an EFS-defining event divided by the number of participants in the efficacy analysis set.
Cohort 6: Rate of Pathologic Responses | At time of surgery (approximately after 3 months treatment)
  Rate of pathologic responses defined as the number of participants with major or complete pathologic response in the surgical specimen from surgery after neo-adjuvant trial treatment divided by the number of participants in the efficacy analysis set.
Cohort 6: ORR at the End of Neo-Adjuvant Treatment (Using RECIST v1.1) | Up to 3 months
  ORR defined as the number of participants with CR or PR as BOR according to response evaluation criteria in solid tumors (RECIST) v1.1 divided by the number of patients in the efficacy analysis set.
Cohort 6: Rate of Progressive Disease at the End of Neo-Adjuvant Treatment (Using RECIST v1.1) | Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (45):
- United States (5):
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Virginia, Fairfax, Virginia
- Australia (4):
  - Scientia Clinical Research, Randwick, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Cancer Research SA, Adelaide, South Australia
  - Monash Health, Clayton, Victoria
- Germany (4):
  - Universitätsklinikum Köln, Cologne
  - Krankenhaus Nordwest GmbH - Institut Fuer Klinisch-Onkologische Forschung (IKF), Frankfurt
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Universitaetsmedizin der Johannes Gutenberg Universitaet Mainz KoeR, Mainz
- Hungary (4):
  - ICON-PRA Budapest, Fázis 1 Vizsgálóhely, Budapest
  - Semmelweis Egyetem ÁOK Belgyógyászati és Onkológiai Klinika, Budapest
  - National Institute of Oncology, Budapest
  - Clinexpert Ltd, Gyöngyös
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Warminsko Mazurskie Centrum Chorob Pluc w Olsztynie, Olsztyn
  - NZOZ Medpolonia Sp. Z o.o, Poznan
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy, Warsaw
- Spain (8):
  - Institut Catala d'Oncologia Badalona, Hospital Germans Trias I Pujol, Badalona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - START Madrid - CIOCC. Grupo Hospital de Madrid (HM) - Centro Integral Oncologico Clara Campal (CIOCC), Madrid
  - Complejo Hospitalario Universitario de Santiago de Compostela (CHUS) - Hospital Clinico Universitario (University Clinical Hospital), Santiago de Compostela
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario y Politecnico La Fe, Valencia
- Turkey (Türkiye) (10):
  - Adana Sehir Hospital, Adana
  - Haceteppe Hospital, Ankara
  - Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara
  - Ankara City Hospital, Ankara
  - Koc University Hospital, Istanbul
  - University Medical Faculty Oncology Institute, Istanbul
  - Yeditepe University, Istanbul
  - Ege University School of Medicine Tulay Aktas Oncology Hospital, Izmir
  - Dokuz Eylul Medical School, Izmir
  - Adana Sehir Hospital, Yüreğir
- United Kingdom (6):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Velindre NHS Trust, Cardiff
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - Guy's and St Thomas NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No